CLINICAL TRIAL: NCT05763589
Title: Study of the Effects of Soy Exposure in Early Life on Bone Development and Gut Microbiota
Status: Active, not recruiting | Type: Observational
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. WONG Man Sau, Professor, The Hong Kong Polytechnic University
Other Study IDs: NTEC-2021-0791
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Child Development
Keywords: Soy isoflavones; Bone development; Soy oligonucleotide; Gut microbiome; Prebiotics; Postbiotics; Early life exposure; Metabolomics; Short-chain fatty acid; Equol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — At around 36-month postpartum, mother and child will provide one urine sample (10-15 ml) for assessing equol production.
  Bone assessment will be performed when the child is at the age of 6 years old in a designated site at the Prince of Wales Hospital in Shatin:
  The child will undergo high-resolution peripheral quantitative computed tomography (HR-pQCT) to measure the cross-sectional geometry, volumetric bone mineral density, and bone microstructure at the distal radius of the non-dominant forearm. The scan region is 4% of the forearm length proximal to the lateral edge of the radial joint surface of the wrist.
  (Optional) The child will provide blood (2-3 ml) and urine sample (10-15 ml) for measuring bone markers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention is involved — No intervention is involved

SUMMARY:
In this project, the investigators aim to investigate the effects of soy consumption at early life on the development of gut microbiota and bone growth. The hypothesis to be tested is that early-life exposure to soy optimize bone growth via the alteration of gut microbiota composition. Clinical samples from mother-child pairs recruited into the SMART Gen Hong Kong cohort will be used to examine the association between maternal soy intake with infant gut microbiota and child's bone development. Primary outcome: Bone mineral density; dynamic bone formation parameters; messenger ribonucleic acid (mRNA) expression of bone markers. Secondary outcome: Gut microbiome profile; metabolomic profile in serum, urine or feces; correlation between soy-induced gut microbiota or metabolites and bone growth. The investigators expect that early life exposure to soy will improve bone growth via gut microbiota and provide scientific evidences for the use of soy preparation in early life as a preventive measure for optimizing bone health.

DETAILED DESCRIPTION:
Peak bone mass, achieved at the end of growth period, plays a critical role in the risk of osteoporotic fractures occurring later in life. A 10% increase in peak bone mass was predicted to delay the development of osteoporosis by 13 years. The determinants of peak bone mass include both genetic (such as gender and race) which accounts for up to 75% of bone mass, and lifestyle factors (such as diet and physical activities) which accounts for the remaining 25%. Lifestyle factors play important roles in optimizing bone accrual during growth, for example, dietary Ca was shown to predict 10-15% of skeletal Ca retention during adolescence while exercise could enhance the effects of dietary Ca via enhancing bone geometry.

Recent studies suggest that gut microbiota is a key regulator of bone mass. Experimental studies showed that bone mineral density (BMD) was altered by ablation of gut microbiota in germ-free mice as well as in mice treated with antibiotics. Moreover, administration of antibiotic either at birth or at weaning was shown to exert a longer-lasting effect on BMD in female C57BL/6 mice at 20 weeks of age but not in male mice. This finding suggests altering microbiota at a critical developmental window has a long-term impact on bone health. Indeed, the establishment of gut microbiota in human is believed to take place beginning at birth in which bacteria from mother will immediately colonize the gastrointestinal (GI) tract of the newborn until its stabilization towards an adult-like configuration during the 3-year period after birth. The development of gut microbiota during this critical period is likely to be affected by different environmental factors, including breastfeeding, diet and antibiotic treatment. Thus, establishing optimal gut microbiota during critical developmental period is a potential mean for enhancing bone health.

The composition of the gut microbiota has been reported to be altered by animal-based diet, Mediterranean diet as well as different dietary factors such as dietary/prebiotic fiber and probiotics. For example, galacto-oligosaccharides is a prebiotic fiber that could increase the proportion of bifidobacteria in GI tract, increase short-chain fatty acids (SCFAs) and decrease cecal pH, thereby increasing mineral absorption, bone biomechanical strength as well as BMD of growing male rats. Similarly, the probiotics Lactobacillus rhamnosus GG was shown to reduce gut permeability, decrease intestinal and bone marrow inflammation, and completely protect against sex steroid-deficiency associated bone loss. The differences in gut microbiota composition is also thought to contribute to the differences in the person's ability to produce equol, a nonsteroidal estrogen metabolized by bacteria from soy isoflavones, that account for the estrogenic actions of soy in bone. Such differences might account for effectiveness of soy isoflavones for protection against bone loss in Asian, but not Western, populations. The ability to produce equol in healthy infants was found to be developmentally regulated and affected by diet composition, in which only trace amounts of equol could be detected in infant plasma at 6 months of age possibly due to the lack of developed gut microflora. Subsequent studies indicate the importance of habitual diets in contributing to equol production in which equol-producers appear to have a higher intake of carbohydrate and dietary fiber, soy and plant protein and lower intake of fat than non-producers. Thus, it is of high importance to identify dietary factors that can optimize the development of gut microbiota and the production of equol for optimizing bone health.

Soy-containing diets are reported to be dietary factors in early life that optimize bone acquisition. Early-life soy exposure was found to promote bone growth and neonatal administration of soy isoflavones could attenuate bone deterioration during adulthood. However, the impact of soy components on gut microbiota in these studies was not characterized, and it is unclear if these bone acquisition effects are related to the actions of soy on gut microbiota composition. Moreover, it should be noted that different soy preparations were being used in different preclinical and clinical studies, including soy isoflavones extract or purified compounds (genistein and daidzein), soy protein isolates with isoflavones, whole soy products (soymilk and other soybean products). The differences in soy preparations might have different effects on the gut microflora, and hence on bone. Indeed, apart from being dietary sources of protein and isoflavones, soybeans are also rich in fibers (polysaccharides and oligosaccharides). Soybean oligosaccharides (SBOS), have been reported to increase the population of bifidobacteria in human fecal samples. In addition, soluble fibers from soy could be fermented by colonic bacteria, leading to SCFAs formation, thereby potentially exerting beneficial effects on bone. Thus, it will be important to identify which dietary components of soy (soy fiber or soy isoflavones) exposed at early life will achieve optimal bone acquisition and gut microbiota.

Alteration of the composition of gut microbiota at early life by dietary soy appears to be a promising approach for enhancing bone growth. However, more studies are needed to address the following questions before any dietary advice for the use of soy in optimizing bone growth can be made: When will be the best time (before birth, nursing or after weaning) for dietary soy exposure for optimal gut microbiota and bone growth? Which component in soy (fiber or isoflavones, or both) offer(s) better effects on bone growth via the modulation of gut microbiome? Which microbes altered by soy are associated with optimal bone growth? Which biomarkers/metabolites (SCFAs, equol, or novel metabolites) can account for the optimal bone growth upon soy exposure?

ELIGIBILITY:
Inclusion Criteria for healthy pregnant women:

1. Chinese mothers aged 18 - 45 years who were in the first trimester of pregnancy
2. Singleton pregnancy
3. Participate voluntarily and capable of giving informed consent

Inclusion Criteria for babies:

The baby of enrolled pregnant women and parents signed written informed consent prior to the initiation of this study.

Exclusion Criteria:

1. Significant medical conditions especially those required long term medications, such as oral steroid, antihypertensive drugs, diabetic medications and lipid-lowering agents, during or before pregnancy
2. History of chronic inflammatory or neoplastic diseases involving the gastrointestinal tract (e.g. inflammatory bowel disease, coeliac disease, colorectal cancer)
3. Significant pregnancy complications, such as intrauterine foetal demise/stillbirth, extreme prematurity, or pre-labour rupture of membranes before 24 weeks
4. Mother with mental incapacity such that they are not able to give informed consent
5. Foetal chromosomal or clinically significant structural abnormalities
6. The current pregnancy is a conception through either sperm or ovum donation

Ages: 3 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: 120 mother-child pairs
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | through study completion, an average of 1 year
  dynamic bone formation parameters; mRNA expression of bone markers

SECONDARY OUTCOMES:
Gut microbiome profile | through study completion, an average of 1 year
  metabolomic profile in serum, urine or feces; correlation between soy-induced gut microbiota or metabolites and bone growth.

CONTACTS AND LOCATIONS:
Overall Officials: Man Sau Wong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, China